CLINICAL TRIAL: NCT05975580
Title: Pharmacotherapy in Conjunction With Lifestyle Counseling for Management of Weight Regain After Bariatric Surgery
Acronym: PROJECT-BARI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kishore M Gadde, MD, Professor In Residence, Surgery, University of California, Irvine
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1849; R01DK129936 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-08-04 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Bariatric surgery; Weight regain; Antiobesity drugs; Treatment of weight regain
MeSH Terms: conditions — Obesity | interventions — Topiramate; Phentermine

STUDY DESIGN:
Intervention Model Description: A total of 120 eligible subjects, with weight regain after bariatric surgery, will be initially randomized in a 3:3:2 ratio to daily treatment with topiramate (TPM) or phentermine (PHEN) or placebo. After 4 months, responders (those with ≥5% weight loss) will continue the same treatment, while nonresponders will be re-randomized to a higher dose of the same drug or phentermine/topiramate combination (PHEN/TPM) during Months 5-12. All randomized subjects will receive lifestyle counseling throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational drugs and placebo capsules will look identical. University of California Irvine Medical Center Investigational Drug Service will dispense the masked study drugs in accordance with randomization. The study statistician who generates the randomization scheme and the research pharmacist who dispenses the study drugs are the only personnel who are unblinded to the randomized assignment. Investigators and all other study personnel and the study subjects will be blinded to the treatment assignment until subjects have completed all visits, all data have been entered, and the data file has been locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group A: Topiramate 50 mg (Experimental): Topiramate will be started at 25 mg daily and the dose will be increased to 50 mg daily after 15 days. Responders at Month 4 will continue the same treatment until Month 12.
  Interventions: Drug: Topiramate
- Group B: Topiramate 100 mg (Experimental): Nonresponders in the topiramate group at Month 4 will be re-randomized in a 1:1 ratio to receive topiramate 100 mg or phentermine/topiramate 15/100 mg during Months 5-12. Doses will be titrated in Month 5.
  Interventions: Drug: Topiramate
- Group C: Phentermine 15 mg/Topiramate 100 mg (Experimental): Nonresponders in the topiramate group at Month 4 will be re-randomized in a 1:1 ratio to receive topiramate 100 mg or phentermine/topiramate 15/100 mg during Months 5-12. Doses will be titrated in Month 5.
  Interventions: Drug: Topiramate; Drug: Phentermine
- Group D: Phentermine 15 mg (Experimental): Phentermine will be started at 7.5 mg daily and the dose will be increased to 15 mg after 15 days. Responders at Month 4 will continue the same treatment until Month 12.
  Interventions: Drug: Phentermine
- Group E: Phentermine 30 mg (Experimental): Nonresponders in the phentermine group at Month 4 will be re-randomized in a 1:1 ratio to receive phentermine 30 mg or phentermine/topiramate 15/100 mg during Months 5-12. Doses will be titrated in Month 5.
  Interventions: Drug: Phentermine
- Group F: Phentermine 15 mg/Topiramate 100 mg (Experimental): Nonresponders in the phentermine group at Month 4 will be re-randomized in a 1:1 ratio to receive phentermine 30 mg or phentermine/topiramate 15/100 mg during Months 5-12. Doses will be titrated in Month 5.
  Interventions: Drug: Topiramate; Drug: Phentermine
- Group P: Placebo (Placebo Comparator): Placebo group will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate is an anticonvulsant (antiepilepsy) drug. IUPAC ID: 2,3:4,5-Bis-O-(1-methylethylidene)-beta-D-fructopyranose sulfamate
  Arms: Group A: Topiramate 50 mg; Group B: Topiramate 100 mg; Group C: Phentermine 15 mg/Topiramate 100 mg; Group F: Phentermine 15 mg/Topiramate 100 mg
Drug: Phentermine — Phentermine belongs to a class of drugs called anorectics, also known as appetite suppressants. IUPAC name 2-methyl-1-phenylpropan-2-amine
  Arms: Group C: Phentermine 15 mg/Topiramate 100 mg; Group D: Phentermine 15 mg; Group E: Phentermine 30 mg; Group F: Phentermine 15 mg/Topiramate 100 mg
Drug: Placebo — Placebo is an inactive substance.
  Arms: Group P: Placebo

SUMMARY:
This is a randomized controlled trial employing a Sequential Multiple Assignment Randomized Trial (SMART) design to test whether pharmacotherapy, in conjunction with lifestyle counseling, can reverse weight regain after bariatric surgery.

DETAILED DESCRIPTION:
Although bariatric surgery is the most effective treatment for severe obesity, a large proportion of patients experience significant weight regain with longer follow-up.

In this randomized controlled trial employing a SMART design, a total of 120 subjects with weight regain after bariatric surgery, will be initially randomized in a 3:3:2 ratio to daily treatment with topiramate (TPM) or phentermine (PHEN) or placebo. After 4 months, responders (those with ≥5% weight loss) will continue the same treatment, while nonresponders will be re-randomized to a higher dose of the same drug or phentermine/topiramate combination (PHEN/TPM) during Months 5-12. All subjects will receive diet and lifestyle counseling throughout the study.

Aim 1: To determine whether pharmacotherapy can reverse post-bariatric surgery weight regain.

Hypothesis: Compared to placebo, all three active drug therapies - TPM, PHEN, and PHEN/TPM will lead to greater percent weight loss at Month 12.

Aim 2: To examine change in energy intake assessed by a dietitian interview.

Hypothesis: Compared to placebo, active drug therapies will lead to greater reduction in energy intake at Month 12.

Aim 3: To examine changes in the most common maladaptive eating behaviors in the post-bariatric surgery patients - grazing, loss-of-control eating, and binge eating.

Hypothesis: Compared to placebo, active drug therapies will lead to decreased maladaptive eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-70 years
2. Had sleeve gastrectomy (SG) or Roux-en-Y gastric bypass (RYGB) at least 18 months ago
3. Weight regain of ≥5% relative to post-surgery nadir weight
4. Body mass index (BMI) ≥30 kg/m2 or ≥27 kg/m2 with weight-related comorbidities
5. Women of childbearing potential must be using appropriate contraception to avoid pregnancy throughout the study, and must have a negative pregnancy test at study entry
6. Must be able to provide written informed consent

Exclusion Criteria:

1. Type 1 diabetes
2. Insulin-dependent type 2 diabetes
3. Fasting plasma glucose (FPG) ≥240 mg/dL
4. Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥150 mm Hg and/or diastolic blood pressure (DBP) ≥100 mm Hg on the average of three seated measurements after being at rest for at least 5 minutes
5. History of significant (as determined by the investigator) and unstable cardiovascular disease including coronary artery disease, arrhythmias, severe congestive heart failure, or stroke
6. Use of monoamine oxidase inhibitors, current or within 2 weeks
7. Hyperthyroidism or other significant thyroid disease
8. Angle-closure glaucoma
9. Agitated states
10. History of drug abuse within the past year
11. Known hypersensitivity or idiosyncrasy to sympathomimetic amines
12. Severe hepatic disease (non-alcoholic fatty liver disease or non-alcoholic steatohepatitis without portal hypertension or cirrhosis is acceptable)
13. End-stage renal disease
14. History of nephrolithiasis
15. Serum triglycerides ≥500 mg/dL
16. Cancer, not in remission, within the past 2 years except for adequately treated basal cell, squamous cell skin cancer, or in-situ cervical cancer
17. History of psychosis or bipolar disorder
18. Suicidal ideation or unstable/untreated major depressive disorder within the past year
19. Use of antidepressant medication that has not been at stable dose for at least 3 months
20. Hospital Anxiety and Depression Scale (HADS) score of ≥11 for depression or anxiety items
21. Binge Eating Scale (BES) score of ≥27
22. Alcohol use disorder within the past year
23. Epilepsy
24. Currently taking phentermine or topiramate or the combination, or products containing these drugs
25. Currently taking stimulants (e.g., Attention Deficit Hyperactivity Disorder medications)
26. Current use of prescription or over-the-counter weight loss drugs or supplements
27. Taking prescription or over-the-counter drugs or products, which in the opinion of the PI, could be associated with significant effects on body weight
28. Planning additional bariatric surgery procedures in the next 13 months
29. History of revisional bariatric surgery (revisional surgery after adjustable gastric banding is acceptable)
30. Currently participating in another weight loss program or have plans to participate in the next 13 months
31. Smoking cessation within the previous 3 months or plans to quit smoking in the next 13 months
32. Pregnant or breastfeeding or planning pregnancy in the coming 13 months
33. History of, or any existing condition that, in the opinion of the Principal Investigator, would interfere with the study outcomes or place the subject at unacceptable risk by participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2027-04-02 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Percent weight loss at Month 12 - Topiramate vs placebo | Month 0, Month 12
  Topiramate (Group 1 [Group A + Group B]) vs placebo (Group P)
Percent weight loss at Month 12 - Phentermine vs placebo | Month 0, Month 12
  Phentermine (Group 2 [Group D + Group E) vs placebo (Group P)
Percent weight loss at Month 12 - Phentermine/Topiramate | Month 0, Month 12
  Phentermine/Topiramate (Group 3 [Group C + Group F]) vs placebo (Group P)

SECONDARY OUTCOMES:
Energy intake | Month 0, Month 12
  Change in energy intake in kcal/d assessed with a dietitian interview. Comparisons between Groups 1, 2, 3 vs placebo.

OTHER OUTCOMES:
Grazing | Months 0, 4, 12
  Change in grazing behavior, assessed with the Grazing Questionnaire. Comparisons between Groups 1, 2, 3 vs placebo.
Loss-of-control eating | Months 0, 4, 12
  Change in loss-of-control eating, assessed with the Loss-of-Control Eating Scale. Comparisons between Groups 1, 2, 3 vs placebo.
Binge eating | Months 0, 4, 12
  Change in binge eating, assessed with the Binge Eating Scale. Comparisons between Groups 1, 2, 3 vs placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore M Gadde, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noria SF, Shelby RD, Atkins KD, Nguyen NT, Gadde KM. Weight Regain After Bariatric Surgery: Scope of the Problem, Causes, Prevention, and Treatment. Curr Diab Rep. 2023 Mar;23(3):31-42. doi: 10.1007/s11892-023-01498-z. Epub 2023 Feb 8. PMID 36752995